CLINICAL TRIAL: NCT07157228
Title: Clinical Characteristics, Etiologies, and Outcomes of Patients With Haematochezia at Al-Rajhi University Hospital.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Rashad Mohamed Mahmoud, residant doctor, Assiut University
Other Study IDs: Haematochezia CP.etiology.out
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Haematochezia
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients >18 years old presenting at the GIT Endoscopy Unit with fresh bleeding per rectum or admitted at Tropical Medicine & Gastroenterology Department, Al-Rajhi University Hospital in a period of one year.

SUMMARY:
Haematochezia is the passage of bright red or maroon blood or blood clots from the rectum, usually originates from a source in lower parts of the gastrointestinal (GI) tract

* In addition, haematochezia can be seen in patients with brisk upper gastrointestinal bleeding (UGIB). The underlying etiology can vary from life threatening variceal bleeding to clinically insignificant haemorrhoidal bleeding . The most common etiology is diverticular bleeding, which accounts for 20% to 55% of cases, followed by intestinal ischemia, inflammatory bowel diseases, anorectal disorders, and neoplasia, which each accounting for around 10% of cases
* LGIB can be mild and intermittent or moderate or severe . Patients with mild bleeding can be electively evaluated as outpatients. While, those with severe bleeding should be hospitalized for management Acute or severe LGIB has an incidence of 20-30 cases/100,000 person years and accounts for 20% of GI bleeds (7-8). The overall mortality rate of LGIB is 2-4% .

Clinical data available at the time of initial patient evaluation can be used to identify patients at high risk for severe bleeding and other adverse outcomes. Several scoring systems have been developed to assess risk in acute LGIB .

To the best of our knowledge, no Egyptian study has addressed the outcome of patients with haematochezia presented at the endoscopy units or has evaluated the clinical utility of risk scores in assessment of patients admitted to hospitals with acute haematochezia. Therefore, we need to study the short-term outcomes of patients with haematochezia (and their predictors) after being managed.

ELIGIBILITY:
Inclusion Criteria:

patients >18 years old presenting at the GIT Endoscopy Unit withfresh bleeding per rectum or admitted at Tropical Medicine & Gastroenterology Department, Al-Rajhi University Hospital in a period of one year.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients with isolated melena without haematochezia.
* Patients who refuse colonoscopy
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients >18 years old presenting at the GIT Endoscopy Unit withfresh bleeding per rectum or admitted at Tropical Medicine & Gastroenterology Department, Al-Rajhi
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
To identify the incidance of haematochezia in patients presented to Al-Rajhi University Hospital. | baseline
  To identify the incidance of haematochezia in patients presented to Al-Rajhi University Hospital.